CLINICAL TRIAL: NCT04890392
Title: A Single-arm Exploratory Study of Safety and Efficacy of Tislelizumab in Combination With S-1 Plus Oxaliplatin as a Neoadjuvant Treatment in Patients With Advanced Gastric/Gastroesophageal Junction Cancer
Brief Title: Tislelizumab Combined With S-1 Plus Oxaliplatin as a Neoadjuvant Treatment in Patients With GC/GEJC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WuhanUHTkx
Record Dates: First submitted 2021-04-27; First posted 2021-05-18 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Advanced Gastric Cancer; Advanced Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 with SOX (Experimental): S-1: 40~60mg Bid，d1~14, q3w Oxaliplatin：130mg/m2，iv drip for 2h，d1, q3w PD-1（Tislelizumab）:200mg,iv drip for at least 1h,d1,q3w
  Interventions: Drug: PD-1 inhibitor(Tislelizumab) ,SOX(S-1+ Oxaliplatin)

INTERVENTIONS:
Drug: PD-1 inhibitor(Tislelizumab) ,SOX(S-1+ Oxaliplatin) — S-1: 40~60mg Bid，d1~14, q3w. Oxaliplatin：130mg/m2，iv drip for 2h，d1, q3w. PD-1（Tislelizumab）:200mg,iv drip for at least 1h,d1,q3w. Stage I: PD1 inhibitor + SOX regimen (q3W) . Stage II: PD1 inhibitor + SOX regimen (q3W) Stage III: PD1 inhibitor + SOX regimen (q3W) . Efficacy evaluation,then followed by surgery.

SUMMARY:
At present, the treatment of advanced gastric/gastroesophageal junction cancer is a research hotspot in the academic community. In Asia, Siewert type II and type III are the main types of advanced gastric/gastroesophageal junction cancer. The current consensus in the academic community for the treatment of this part of the tumor is based on the principles of diagnosis and treatment of gastric cancer, of which the value of neoadjuvant therapy in this part of the tumor has been paid more and more attention by scholars. However, there is no highly recognized neoadjuvant therapy. The current situation will promote the development of advanced gastric/gastroesophageal junction cancer to accurate preoperative staging, more accurate population screening, more accurate targets and molecular markers. Immunotherapy is a promising application in oncology. Several PD1/PD-L1 monoclonal antibodies are approved by FDA for the clinical treatment of melanoma and other tumors. Previous clinical studies have shown that PD1/PD-L1 has limited efficacy in digestive tract tumors. However, on ASCO in 2020, Asian analysis of KEYNOTE-062 study showed that in HER-2 negative advanced gastric cancer with PD-1 combined positive score (CPS) ≥ 1 and CPS ≥ 10, the OS of PD-1 inhibitor treatment was superior to that of chemotherapy group, with 24-month OS rate (CPS ≥ 1, 45% VS 23%, CPS ≥ 10, 54% VS 27%). Meanwhile, the results of PACIFIC study phase III clinical trial showed that the 3-year OS of PD-L1 monoclonal antibody combined with radiotherapy in advanced unresectable lung cancer was as high as 57%, which is expected to completely rewrite its clinical practice. Immunotherapy is promising in cancer therapy. This study intends to use immunotherapy combined with SOX (S-1 + Oxaliplatin) as a neoadjuvant therapy for advanced gastric/gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Obtaining written informed consent from patient in advance.
2. Gastroscopy confirmed adenocarcinoma of the gastroesophageal junction or stomach and biopsy pathology confirmed adenocarcinoma of the stomach.
3. ECOG 0-1
4. Normal function of major organs, meeting the following criteria:

   Blood routine test criteria should be met (Patients for 14 days were not transfused with blood products and not corrected with G-CSF and other hematopoietic stimulating factors)
   1. HB≥90 g/L；
   2. ANC≥1.5×10^9/L；
   3. PLT≥125×10^9/L；

   Chemistry panel meeting the following criteria:
   1. TBIL< 1.5ULN;
   2. ALT and AST< 2.5ULN, but< 5ULN for patients with liver metastasis;
   3. serum Cr ≤ 1.25ULN or endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula);
5. Women of childbearing potential must have used reliable contraception or had a pregnancy test (serum or urine) within 7 days prior to enrollment and had a negative result, and be willing to use an appropriate method of contraception during the trial and for 8 weeks after administration of the trial drug. For men, agree to use an appropriate method of contraception or have been surgically sterilized during the trial and for 8 weeks after receiving study drug.
6. Advanced gastric cancer as assessed by ultrasonography and/or gastric CT (cT3-T4a, N+, M0).

Exclusion Criteria:

1. Peritoneal dissemination
2. Patients who previously received platinum, fluoropyrimidine chemotherapy or targeted therapy, and patients who received radiotherapy to target lesion during combined therapy
3. Multiple factors affecting oral medications (e.g., inability to swallow, chronic diarrhea, bowel obstruction, etc.)
4. History of melena or hematemesis in the past three months, or patients with high-risk bleeding such as intestinal perforation, gastric perforation, large area ulcer, or patients with active digestive ulcer lesions in the stomach and fecal occult blood (+ +).
5. Patients with hypertension and uncontrolled by antihypertensive treatment alone (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg); patients with a history of unstable angina; patients newly diagnosed as angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; arrhythmia (including QT ≥ 450 ms for men, ≥ 470 ms for women) requiring long-term use of antiarrhythmic drugs and New York Heart Association class ≥ II cardiac insufficiency; Doppler ultrasound assessment: ejection fraction (LVEF) < 50%.
6. Urine routine showed urine protein ≥(+ +)and confirmed 24-hour urine protein >1.0g
7. Long-term unhealed wounds or incompletely healed fractures
8. Patients with abnormal coagulation function and bleeding tendency (the following criteria must be met within 14 days before enrollment: INR is within normal range without anticoagulant); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; patients treated with low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (the daily dose does not exceed 100 mg) for preventive purposes are allowed under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5
9. Hyperactive/venous thrombotic events within 1 year before screening, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis (except venous thrombosis caused by previous chemotherapy that has been cured by the investigator) and pulmonary embolism
10. Patients with a history of psychotropic substance abuse who cannot quit or have mental disorders
11. Patients with concomitant diseases that seriously jeopardize the patient's safety or affect the patient's completion of the study as judged by the investigator
12. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-01-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 years
  Defined as the proportion of patients whose tumors shrink for a certain period of time

SECONDARY OUTCOMES:
Disease control rate (DCR) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 years
  Defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time
pCR rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Pathological complete response
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
postoperative complications | Investigator assessment,from the initiation date of the operation day, assessed up to 1 years.
  Complications refer to the occurrence of another or several diseases related to the therapeutic behavior of this disease during the treatment of a certain disease

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College of HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yin Y, Lin Y, Yang M, Lv J, Liu J, Wu K, Liu K, Li A, Shuai X, Cai K, Wang Z, Wang G, Shen J, Zhang P, Tao K. Neoadjuvant tislelizumab and tegafur/gimeracil/octeracil (S-1) plus oxaliplatin in patients with locally advanced gastric or gastroesophageal junction cancer: Early results of a phase 2, single-arm trial. Front Oncol. 2022 Aug 30;12:959295. doi: 10.3389/fonc.2022.959295. eCollection 2022. PMID 36158692